CLINICAL TRIAL: NCT06791356
Title: Cognitive Behavioral Therapy for Insomnia in Older African American Adults
Brief Title: CBT-I in Older African American Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mark A. Gluck, PhD, Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2024000293; 1R01AG078211 (NIH)
Record Dates: First submitted 2025-01-10; First posted 2025-01-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Older Adults (65 Years and Older)
Keywords: insomnia; cognitive-behavioral therapy for insomnia; African Americans
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I (Experimental)
  Interventions: Behavioral: Cognitive-behavioral therapy for insomnia
- Sleep hygiene education (Active Comparator)
  Interventions: Behavioral: Sleep hygiene education

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy for insomnia — 8 sessions of therapy that focus on psychoeducation about sleep hygiene, cognitive restructuring of dysfunctional beliefs that reinforce insomnia, stimulus control to eliminate the association between the bed and wakefulness, sleep restriction in order to establish a consistent sleep schedule, and relaxation training to reduce anxiety that interferes with sleep
  Arms: CBT-I
Behavioral: Sleep hygiene education — One session of education about behavioral strategies to optimize sleep quality
  Arms: Sleep hygiene education

SUMMARY:
Sleep problems, like insomnia, are common in older African Americans. About 25% of older adults in the US have at least 2 symptoms of insomnia, such as having trouble falling asleep, staying asleep, or getting good sleep for a month or more. Cognitive Behavioral Therapy for Insomnia (CBT-I) is a recommended non-pharmacological treatment for insomnia. Unlike medicines that might only help for a short time or have many side effects, CBT-I deals with the root causes of insomnia. It helps people change how they think and act about sleep, leading to better habits and attitudes. This can make sleep better for a long time, even after the treatment is over. While CBT-I is commonly used among adults with insomnia, its benefits among older adults and specifically older African American adults are not well understood. Thus, the current pilot study will investigate the feasibility of CBT-I in older African American adults and establish preliminary evidence for the potential benefit of CBT-I on sleep as well as cognition in this population.

For this study, participants will be asked to complete pencil-and-paper questionnaires, psychological tests of cognition, 7-day actigraphy, 2 nights of at home sleep monitoring, which collects specific sleep measures such as brain waves and sleep stage timing, and computer-based neuropsychological tests before and after intervention. Study interventions will consist of 8 weekly sleep training sessions via Zoom or a single session of education on strategies to improve sleep quality. Sleep training sessions will include education about strategies to improve sleep quality, changing thought process that contribute to insomnia, training the brain on the optimal sleep environment, and reducing sleep initially to establish a consistent sleep schedule before increasing sleep time. Three months after the post-intervention visit, participants will be asked to come back in for a follow-up evaluation which consists of complete pencil-and-paper questionnaires, psychological tests of cognition, 7-day actigraphy, 2 nights of at home sleep monitoring, and computer-based neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

* Reading level 6th grade or better and can speak and understand English well.
* Self-identify as African American or Black.
* Ages 60 and over.
* Score of >2 in PSQI sleep duration, sleep disturbance, or overall sleep quality calculated components.
* Participating in the "Pathways to Healthy Aging in African Americans" study.
* Has established chronic insomnia issues for at least three months.
* Subjects must be willing to participate in 8 sessions of CBT-I via Zoom for the CBT-I group.
* Subjects must be willing to come for pre/post assessment visits.
* MoCA score of between 20-26.

Exclusion Criteria:

* Currently taking any of the following medications consistently: Benzodiazepines (ProSom, Restoril, Ativan and Xanax); Z Drugs (eszopiclone (Lunesta), zaleplon (Sonata) and zolpidem (Ambien, Ambien CR, Edluar, and Zolpimist); antidepressants that affect sleep (doxepin, mirtazapine, trazodone); antihistamines (diphenhydramine and doxylamine succinate); barbiturates (methohexital, pentobarbital, primidone, secobarbital).
* Diagnosed with any sleep disorder other than insomnia (i.e. obstructive sleep apnea using STOP-BANG, restless leg syndrome, REM sleep behavior disorder, etc.).
* Classified as high fall risk.
* Primary causes for frequent awakenings are due to a medical condition that is not related to insomnia, such as chronic pain, urinary frequency, upper respiratory infection.
* Previous experience with CBT-I.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Adherence | From enrollment to the end of treatment at 8 weeks
  Number of sessions completed, sleep diary completion rate

SECONDARY OUTCOMES:
Sleep efficiency - immediate treatment effect | From enrollment to the end of treatment at 8 weeks
  Ratio of number of hours actually slept over total time in bed
Cognitive task performance - immediate treatment effect | From enrollment to the end of treatment at 8 weeks
  Performance in Rutgers Acquired Equivalence (generalization) task

OTHER OUTCOMES:
Sleep efficiency - longer-term treatment effect | 12 weeks after end of treatment
  Ratio of number of hours actually slept over total time in bed
Cognitive task performance - longer-term treatment effect | 12 weeks after end of treatment
  Performance in Rutgers Acquired Equivalence (generalization) task

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gluck, PhD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No